CLINICAL TRIAL: NCT02738112
Title: Hyoid Suspension to the Mandible for the Treatment of Obstructive Sleep Apnea
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Abidin, Michael, M.D. (Individual)
Responsible Party: Sponsor
Other Study IDs: HS 2016.0
Record Dates: First submitted 2016-04-11; First posted 2016-04-14 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Encore System — Hyo-mandibular suspension

SUMMARY:
Hyo-mandibular suspension has been previously studied as a treatment for obstructive sleep apnea (OSA) and has shown to be highly effective.

This is a prospective, multi-center, registry during which 30 subjects with OSA will be considered for hyo-mandubular suspension treatment. After obtaining informed consent and meeting all inclusions and exclusion criteria, subjects will be treated using the Encore System. Subject follow-up with the physician or nurse will occur at one (1) week, one (1) month, three (3) months, and twelve (12) months.

This study will assess the effectiveness of hyoid suspension in reducing the apnea-hypopnea index (AHI), and improving the Epworth Sleepiness Scale (ESS), snoring (VAS) and functional outcome (FOSQ) for the treatment of obstructive sleep apnea (OSA). In addition, the study will evaluate the effect that the change in hyoid position has on the airway anatomy.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) has become a major heath problem in the United States. With prevalence in middle-aged adults of 2 to 4% of the population, untreated OSA has been implicated in increased risk for cardiovascular disease, including hypertension and heart failure.

The first line and most common treatment for OSA is continuous positive airway pressure (CPAP) treatment, utilized by an estimated 3 million Americans. CPAP is effective in reducing the AHI if used properly. However, the nasal mask required for CPAP during sleep leads to poor acceptance and compliance rates. Published studies on CPAP have shown that only 58 to 80% of patients accept CPAP therapy,, and further 65 to 90% of these patients exhibit long-term compliance with CPAP. Additionally, there are many patients who would choose other therapy besides CPAP.

Patients cite a number of issues with CPAP, namely discomfort and inability to sleep while connected to an air pump. Auto-titrating CPAP, heated and humidified air, and bi-PAP (different pressures on inspiration and expiration) have improved patient compliance, but there remains a significant unmet clinical need.

It is widely accepted that the region behind the tongue is a major site of collapse during obstructive sleep apnea. In fact, there are many surgical procedures performed currently to address tongue base collapse. These include: RF ablation (Somnoplasty) of the tongue base; genioglossus advancement; Medtronic's Repose system for tongue base suspension; hyoid suspension; and maxillomandibular advancement (MMA). The change in airway dimension after MMA surgery on the lateral cephalograph is presented in Figure 1.

One of the principal mechanisms of effect of MMA surgery is to move the base of the tongue and the attached structures forward. Hyo-mandibular suspension has been previously studied as a treatment for OSA and has shown to be highly effective.

This is a prospective, multi-center, registry during which 30 subjects with OSA will be considered for hyo-mandubular suspension treatment. After obtaining informed consent and meeting all inclusions and exclusion criteria, subjects will be treated using the Encore System. Subject follow-up with the physician or nurse will occur at one (1) week, one (1) month, three (3) months, and twelve (12) months.

This study will assess the effectiveness of hyoid suspension in reducing the apnea-hypopnea index (AHI), and improving the Epworth Sleepiness Scale (ESS), snoring (VAS) and functional outcome (FOSQ) for the treatment of obstructive sleep apnea (OSA). In addition, the study will evaluate the effect that the change in hyoid position has on the airway anatomy.

ELIGIBILITY:
Inclusion Criteria:

1. Documented diagnosis of moderate or severe obstructive sleep apnea (AHI between 20 and 60/hour) evaluated with a sleep study within 12 months prior to the planned procedure
2. Age ≥ 20 and ≤ 65 years old
3. Body Mass Index (BMI) ≤ 36 (kg/m2)
4. Patient has been offered CPAP and has refused or failed to continue CPAP treatment or is noncompliant with CPAP
5. Significant airway narrowing while mild posterior is pressure applied to hyoid bone
6. Evidence of hypopharyngeal obstruction via pharyngoscopy
7. Signed informed consent to participate in this clinical study

Exclusion Criteria:

Patient History

1. Prior OSA surgery (uvulopalatopharyngoplasty [UPPP], tonsillectomy and nasal surgery are acceptable)
2. Active systemic infection
3. Allergy to any medication used during implantation
4. Previous history of neck or upper respiratory tract cancer
5. Radiation therapy to neck or upper respiratory tract
6. Significant dysphagia or speech disorder Anatomical Considerations

1. Identified obvious palatal stenosis 2. Enlarged tonsils (3+) 3. Anatomy unable to accommodate the implant

Other

1. Other medical, social or psychological problems that, in the opinion of the investigator, preclude patient from receiving this treatment, as well as the procedures and evaluations pre- and post-treatment
2. Enrollment in another pharmacological or medical device study that may effect or bias the results of this clinical study
3. Unable and/or not willing to comply with treatment follow-up requirements
4. Pregnancy (Female subjects of childbearing potential must have a negative pregnancy test prior to enrollment.)
5. Lack of insurance coverage for procedure and PSG follow up and unwillingness to self pay
6. Unwilling or unable to give signed informed consent

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with obstructive sleep apnea (OSA) who meet the inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-03 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index (AHI) | 3 months

SECONDARY OUTCOMES:
Hyoid position and airway dimension measurement | 3 months
Functional Outcomes of Sleep Questionnaire (FOSQ) | 3 months
Snoring Scale (Visual Acuity Scale) | 3 months
Epworth Sleeping Scale | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Abidin, MD, Principal Investigator — Private Practice
Locations (1):
- Michael Abidin, Alexandria, Virginia, United States

IPD SHARING:
Plan to Share IPD: No